CLINICAL TRIAL: NCT06947720
Title: Research on Ultrasound Diagnostic Criteria for Intracranial and Extracranial Arterial Serial Stenosis
Status: Not yet recruiting | Type: Observational
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Other Study IDs: xwzc202500203
Record Dates: First submitted 2025-04-20; First posted 2025-04-27 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Ischemic Stroke; Carotid Stenosis
Keywords: Serial stenosis; hemodynamics; Ultrasound diagnostic criteria; prediction model
MeSH Terms: conditions — Ischemic Stroke; Carotid Stenosis | interventions — Stents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (10):
- Mild stenosis group without collateral circulation: There is no anterior communicating artery, posterior communicating artery, or internal external carotid artery in the skull, and the degree of stenosis in the V4 segment of the middle cerebral artery or vertebral artery is less than 50%
  Interventions: Procedure: stenting
- Group without collateral circulation and stenosis: There is no anterior communicating artery, posterior communicating artery, or internal carotid external artery in the skull, and there is no stenosis in the V4 segment of the affected middle cerebral artery or vertebral artery.
  Interventions: Procedure: stenting
- Moderate stenosis group without collateral circulation: There is no anterior communicating artery, posterior communicating artery, or internal carotid external artery in the skull, and the degree of stenosis in the V4 segment of the affected middle cerebral artery or vertebral artery is 50-69%.
  Interventions: Procedure: stenting
- Severe stenosis group without collateral circulation: There is no anterior communicating artery, posterior communicating artery, or internal carotid external artery in the skull, and the degree of stenosis in the V4 segment of the affected middle cerebral artery or vertebral artery is 70-99%.
  Interventions: Procedure: stenting
- Group with collateral circulation and no stenosis: There are anterior or posterior communicating arteries or internal external carotid arteries in the skull, and there is no stenosis in the V4 segment of the affected middle cerebral artery or vertebral artery.
  Interventions: Procedure: stenting
- Mild stenosis of collateral circulation group: There are anterior or posterior communicating arteries or internal external carotid arteries in the skull, and the degree of stenosis in the V4 segment of the affected middle cerebral artery or vertebral artery is less than 50%.
  Interventions: Procedure: stenting
- Moderate stenosis of collateral circulation group: There are anterior or posterior communicating arteries or internal external carotid arteries in the skull, and the degree of stenosis in the V4 segment of the affected middle cerebral artery or vertebral artery is 50-69%.
  Interventions: Procedure: stenting
- Group with severe stenosis of collateral circulation: There are anterior or posterior communicating arteries or internal external carotid arteries in the skull, and the degree of stenosis in the V4 segment of the affected middle cerebral artery or vertebral artery is 70-99%.
  Interventions: Procedure: stenting
- End event group: During the 1-year follow-up after surgery, the patient experienced new stroke events such as ischemic stroke, transient ischemic attack, and hemorrhagic stroke.
  Interventions: Procedure: stenting
- Group without endpoint events: At the 1-year follow-up after surgery, the patient did not experience any new stroke events such as ischemic stroke, transient ischemic attack, or hemorrhagic stroke.
  Interventions: Procedure: stenting

INTERVENTIONS:
Procedure: stenting — All individuals are anesthetized, with local or general anesthesia depending on the patient's level of cooperation. During the surgery, heparin must be injected intravenously to control the activated clotting time between 250-300 seconds. The surgery is performed via the femoral artery, and the choice of stent type and size, as well as any required equipment, are determined by the intervention personnel themselves.

SUMMARY:
This study utilized different hemodynamic parameters of transcranial color-coded Doppler (TCCD) and transcranial Doppler (TCD) to conduct ultrasonic grading evaluation on middle cerebral artery (MCA) stenosis severity in patients with severe extracranial internal carotid artery stenosis, as well as intracranial V4 segment stenosis severity in patients with severe vertebral artery (VA) origin stenosis. The aim was to establish ultrasonic diagnostic criteria and provide reference basis for clinical treatment decision-making. Clarify the distribution of stroke risk factors, establish and evaluate stroke risk identification and prediction models. Patient cohort: Individuals undergoing carotid artery stenting or vertebral artery stenting, including those with either 1) severe extracranial internal carotid artery stenosis combined with ipsilateral MCA tandem stenosis, or 2) unilateral severe vertebral artery origin stenosis combined with intracranial V4 segment tandem stenosis. Collected data included demographic information, vascular ultrasound findings, and imaging examination results. All patients underwent a 1-year follow-up investigation documenting follow-up vascular ultrasound results, laboratory test results, imaging findings, clinical symptoms (ischemic stroke, transient ischemic attack, hemorrhagic stroke), and occurrence of endpoint events.

DETAILED DESCRIPTION:
This study retrospectively and consecutively enrolled 700 patients diagnosed with either 1) severe extracranial internal carotid artery stenosis combined with ipsilateral middle cerebral artery (MCA) tandem stenosis, or 2) unilateral severe vertebral artery (VA) origin stenosis combined with intracranial V4 segment tandem stenosis, who underwent carotid artery stenting or vertebral artery stenting at our institution. Demographic information, vascular ultrasound findings, and imaging examination results were collected and recorded. All enrolled patients underwent a 1-year follow-up investigation. Follow-up data included vascular ultrasound results, laboratory test results, imaging findings, clinical symptoms (ischemic stroke, transient ischemic attack, hemorrhagic stroke), and documentation of endpoint events. The primary endpoint was the 12-month incidence of new-onset stroke events, defined as ischemic stroke, transient ischemic attack, or hemorrhagic stroke.

The study utilized transcranial color-coded Doppler (TCCD) and transcranial Doppler (TCD) hemodynamic parameters to ultrasonically grade MCA stenosis severity in patients with severe extracranial internal carotid artery stenosis and intracranial V4 segment stenosis severity in patients with severe VA origin stenosis. The goal was to establish ultrasound diagnostic criteria and provide a reference basis for clinical treatment decision-making. Additionally, the distribution of stroke risk factors was analyzed, and a risk identification and prediction model for stroke was developed and evaluated.

Patients were first stratified into two groups based on the presence or absence of collateral circulation. Further subgroup classification was performed according to the degree of MCA stenosis (on digital subtraction angiography [DSA]) or V4 segment stenosis: no stenosis, mild stenosis, moderate stenosis, and severe stenosis. Finally, patients were categorized into either the endpoint event group or the non-event group based on the occurrence of endpoint events during follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed by carotid ultrasound with severe stenosis of the extracranial segment of the internal carotid artery or severe stenosis of the initial segment of the unilateral vertebral artery;
2. Perform stent placement surgery within 2 weeks of ultrasound examination, and perform DSA and CTA examinations;
3. Age ≥ 18 years old;
4. Clinical data is complete.

Exclusion Criteria:

1. Bilateral temporal windows are not transparent to sound;
2. Patients with severe stenosis of the extracranial segment of the internal carotid artery have ipsilateral MCA occlusion/ipsilateral common carotid artery severe stenosis or occlusion;
3. Patients with severe stenosis of the extracranial segment of the internal carotid artery have severe stenosis of the contralateral carotid artery;
4. Patients with severe stenosis or occlusion of the anterior circulation in the initial segment of unilateral vertebral artery;
5. Severe stenosis or occlusion of bilateral subclavian arteries;
6. Vasospasm caused by subarachnoid hemorrhage, etc;
7. Related MCA or vertebral artery thrombolysis or endovascular treatment;
8. Arrhythmias such as atrial fibrillation or heart failure that affect velocity measurement;
9. CT, MRI, DSA examination contraindications or refusal of examination;
10. Severe bleeding disorders or coagulation dysfunction;
11. Merge serious diseases of other organs or tissues.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female patients over 18 years old with severe stenosis of the extracranial segment of the internal carotid artery or severe stenosis of the initial segment of the unilateral vertebral artery, who undergo carotid or vertebral artery stenting
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Ultrasound diagnostic criteria for serial stenosis | From preoperative TCCD assessment to surgical completion
  Ultrasound standards for assessing the degree of stenosis in the ipsilateral middle cerebral artery or vertebral artery V4 segment in patients with severe stenosis of the extracranial segment of the internal carotid artery or the initial segment of the vertebral artery, using different hemodynamic parameters
The occurrence of the endpoint event | Within 1 year after surgery
  At the 1-year follow-up after surgery, whether ischemic stroke, transient ischemic attack, and hemorrhagic stroke occurred.

CONTACTS AND LOCATIONS:
Overall Officials: Yingqi Xing, Principal Investigator — Vascular Ultrasound Diagnosis Department, Xuanwu Hospital
Locations (1):
- Department of Vascular Ultrasound, Xuanwu Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Du B, Wong EH, Jiang WJ. Long-term outcome of tandem stenting for stenoses of the intracranial vertebrobasilar artery and vertebral ostium. AJNR Am J Neuroradiol. 2009 Apr;30(4):840-4. doi: 10.3174/ajnr.A1427. Epub 2009 Mar 11. PMID 19279273
- [Background] Ballotta E, Toniato A, Da Roit A, Baracchini C. Clinical Outcomes of Carotid Endarterectomy in Symptomatic and Asymptomatic Patients with Ipsilateral Intracranial Stenosis. World J Surg. 2015 Nov;39(11):2823-30. doi: 10.1007/s00268-015-3165-7. PMID 26243559
- [Background] Ryu JC, Lee SH, Yoo JS, Kwon B, Song Y, Lee DH, Bae JH, Chang JY, Kang DW, Kwon SU, Kim JS, Kim BJ. Prognosis of Proximal and Distal Vertebrobasilar Artery Stent Placement. AJNR Am J Neuroradiol. 2024 Nov 7;45(11):1685-1691. doi: 10.3174/ajnr.A8389. PMID 39389775
- [Background] Zhang J, Xing Y, Cui L. Duplex Ultrasonography for the Evaluation of Extracranial Vertebral Artery: A Prospective Comparison With Digital Subtraction Angiography. Front Neurol. 2022 Jun 27;13:814972. doi: 10.3389/fneur.2022.814972. eCollection 2022. PMID 35832174
- [Background] Liu S, Huang ZL, Sun YR, Liu L, Qi H, Wei LY. Application value of transcranial contrast-enhanced ultrasonography in evaluating middle cerebral artery stenosis. Eur Rev Med Pharmacol Sci. 2023 Jan;27(1):224-232. doi: 10.26355/eurrev_202301_30875. PMID 36647872